CLINICAL TRIAL: NCT00235105
Title: Adalimumab in Early Axial Spondyloarthritis (Without Radiological Sacroiliitis): Placebo Controlled Phase Over 3 Months Followed by a 9 Months Open Extension Phase
Brief Title: D2E7-Early AS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Abbott (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A01
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-10

CONDITIONS: Ankylosing Spondylitis
Keywords: early ankylosing spondylitis; spondyloarthritis; trial; adalimumab
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab 40 mg sc every other week

SUMMARY:
Reduction of signs and symptoms in patients with moderate to severely early axial spondyloarthritis (without radiological sacroiliitis) who have had an inadequate response to or do not tolerate NSAID therapy.

Study Objectives:Efficacy -To assess whether patients with moderate to severely active early axial spondyloarthritis (without radiological sacroiliitis) will show response when adalimumab is added to the pre-existing or in case of intolerance to NSAID therapy. Response will be measured at week 12 by change of efficacy parameters compared to baseline.Safety - To demonstrate the safety of adalimumab in study patients with moderate to severely active early axial spondyloarthritis (without radiological sacroiliitis) in patients who have had an inadequate response to or do not tolerate NSAID therapy.

DETAILED DESCRIPTION:
The study is a two center 12-week double-blind, placebo-controlled trial of adalimumab in patients with moderate to severely active axial spondyloarthritis (without radiological sacroiliitis) who have had an inadequate response to who are or intolerant to NSAID therapy. Patients may have been treated in the past with concomitant DMARDs. For these patients a washout period of at least 4 weeks is necessary. If Leflunomide was discontinued, it should be stopped at least 3 months or should be washed out within 4 weeks before study start. Patients who have been treated previously with approved biologics are allowed to enter the study if they failed due to lack of efficacy and/or intolerance. The placebo-controlled treatment period of 12 weeks will be followed by an open-label maintenance therapy up to Week 52. Following screening and baseline evaluations, patients will be assessed at Weeks 2, 4, 8, and 12. During the maintenance therapy visits will be performed at Weeks 16, 20 and every eight weeks thereafter.Efficacy and safety measurements will be recorded throughout the entire 52 weeks study.Non-responders (fail to reach ASAS 40) at and after week 12 of open label therapy (at week 24), will be eligible for adalimumab dose escalation to 40 mg weekly.The study will be followed by a 24 weeks follow up phase. During this period the patients will be assessed every eight weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years of age or older who have moderate to severely active axial spondyloarthritis.

Diagnosis made by:Chronic low back pain (duration > 3 months, onset < 50 years of age)plus 3 out of the 6 following criteria (including two of the following three criteria: inflammatory back pain, positive for HLA-B27 and positive MRI showing acute inflammatory lesions in spine or ISG)

* Inflammatory back pain1
* Good or very good response to NSAIDs
* One or more of the following extraspinal manifestations: uveitis, peripheral arthritis, enthesitis
* HLA-B27 positive
* Positive MRI showing acute inflammatory lesions in spine or ISG
* Positive family history for SpA Active disease is defined as a BASDAI score of equal or more than 4, back pain score (BASDAI question 2) of equal or more than 4 despite concurrent NSAID therapy, or intolerance to NSAIDs.

Other inclusion criteria include:

If on prednisone, equal or less than 7.5 mg per day; stable for 4 weeks prior to baseline.

An evaluation for latent tuberculosis infection will be performed using a Mendel Mantoux Test with 10TE (PPD), reading a chest x-ray, which should have been performed within the last 12 weeks before inclusion, and history of exposure to infected subjects. Patients who have evidence of latent TB infection should be given prophylaxis in accordance with local guidelines (Isoniazid 300 mg with adequate substitution of vitamin B6 for 9 months or 600 mg Rifampicine for 6 months). The prophylaxis will start 4 weeks before adalimumab is administered. After 2 weeks of prophylaxis blood tests (liver enzymes, creatinine and blood count) will be obtained. Patients with documented prophylaxis in the past need not to repeat this treatment.

Women of child bearing potential must have a negative pregnancy test at study baseline and use an adequate method of contraception (including 3 months after study completion). Sexual active men must use an accepted method of contraception including 3 months after study completion.

Able to self-administer injectable drug supplies or have a caregiver who will do so.

Able to store injectable test article at 2° to 8° C.

Exclusion Criteria:

Definite ankylosing spondylitis (according to modified New York criteria, sacroiliitis ³ grade 2 bilaterally or grade 3 to 4 unilaterally) History of active tuberculosis (TB), histoplasmosis or listeriosis. History of positive HIV status. Positive serology for hepatitis B or C indicating active infection, in case of hepatitis B also if indicating chronic infection History of malignancy other than carcinoma in situ of the cervix or adequately treated non-metastatic squamous or basal cell skin carcinoma.

Antibiotic treatment within 3 weeks prior to screening. Treatment with biologicals within the last 12 weeks If on DMARDs a washout period of at least 4 weeks is necessary. If Leflunomide was discontinued, it should be stopped at least 3 months or should be washed out within 4 weeks before study start.

History of uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke (within 3 months), ongoing congestive heart failure, and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.

Female subjects who are pregnant or breast-feeding. Previous diagnosis or signs of demyelinating diseases History of systemic lupus erythematosusReceipt of any live (attenuated) vaccines within 4 weeks before screening visit Laboratory exclusions are: hemoglobin level < 8,5 mg/dl, white blood cell count < 3.5 x109/l, platelet count < 125 x 109 /l, creatinine level > 175 µmol/liver enzymes or alkaline phosphatase >2 times the upper limit of normal.

Participation in trials of other investigational medications within 30 days of entering the study Clinical examination showing significant abnormalities of clinical relevance History or current evidence of abuse of "hard" drugs (e.g. cocaine/heroine) or alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2005-03; Study Completion 2007-06

PRIMARY OUTCOMES:
ASAS 40 at week 12

SECONDARY OUTCOMES:
ASAS 20, 70·
BASDAI 20, 50, 70
BASFI (absolute change from Baseline)
Mobility examinations: BASMI, Chest Wall Expansion
DC-ART20 (5 out of 6)
CRP, ESR
Quality of Life: SF-36
Numeric Rating Scale (NRS) - physicians global, patients global, general pain, nocturnal pain
Enthesitis index (Maastricht scale)
swollen joint count
EQ-5D
Safety Evaluations: Adverse events, vital signs, physical examination results, and clinical laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, Prof., Principal Investigator — Charité Campus Benjamin Franklin, Rheumatology
Locations (2):
- Germany (2):
  - Charité Campus Benjamin Franklin, Rheumatology, Berlin
  - Rheumazentrum Ruhrgebiet, Herne

REFERENCES:
- [Derived] Weiss A, Song IH, Haibel H, Listing J, Sieper J. Good correlation between changes in objective and subjective signs of inflammation in patients with short- but not long duration of axial spondyloarthritis treated with tumor necrosis factor-blockers. Arthritis Res Ther. 2014 Jan 30;16(1):R35. doi: 10.1186/ar4464. PMID 24476416
- [Derived] Haibel H, Heldmann F, Braun J, Listing J, Kupper H, Sieper J. Long-term efficacy of adalimumab after drug withdrawal and retreatment in patients with active non-radiographically evident axial spondyloarthritis who experience a flare. Arthritis Rheum. 2013 Aug;65(8):2211-3. doi: 10.1002/art.38014. No abstract available. PMID 23686466
- [Derived] Haibel H, Rudwaleit M, Listing J, Heldmann F, Wong RL, Kupper H, Braun J, Sieper J. Efficacy of adalimumab in the treatment of axial spondylarthritis without radiographically defined sacroiliitis: results of a twelve-week randomized, double-blind, placebo-controlled trial followed by an open-label extension up to week fifty-two. Arthritis Rheum. 2008 Jul;58(7):1981-91. doi: 10.1002/art.23606. PMID 18576337